CLINICAL TRIAL: NCT04035798
Title: The Potential Therapeutic Effects of add-on Low Dose Memantine to Improve Cognitive Deficits in Middle-to-old Aged Bipolar II Disorder Patients
Brief Title: add-on Low Dose Memantine in Middle-to-old Aged Bipolar II Disorder Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Tzu-Yun Wang, Principal Investigator, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-BR-107-095
Record Dates: First submitted 2019-07-01; First posted 2019-07-29 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Bipolar II Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- memantine (MM) (Experimental): The participants will receive memantine 5mg (1 capsule) per day for 12 weeks.
  Interventions: Drug: Memantine or placebo
- Placebo (Placebo Comparator): The participants will receive one capsule of placebo per day for 12 weeks.
  Interventions: Drug: Memantine or placebo

INTERVENTIONS:
Drug: Memantine or placebo — BP-II patients who are older than 40 years old will be recruited, and allocate them to add-on memantine or placebo plus standard valproic acid treatment in a 1: 1 ratio. The participants will receive memantine 5mg/day or placebo treatment for 12 weeks.

SUMMARY:
The investigators hypothesized that add-on memantine (MM) 5 mg/day may reduce chronic inflammation, and subsequently improve neuro-progression process and cognitive function in middle-to-old aged bipolar II disorder (BP-II) patients. In current proposal, the investigators will conduct a randomized double-blind placebo-controlled study. The investigators will recruit 100-120 patients with BP-II who are older than 40 years old in three years, and allocate them to add-on MM or placebo plus standard valproic acid treatment in a 1: 1 ratio. The investigators will follow up the participants for 12 weeks and measure the severity of mood symptoms, neuropsychological tests and inflammatory markers to evaluate the therapeutic effects of add-on MM.

DETAILED DESCRIPTION:
Emerging evidence showed that chronic inflammation and neuro-progression underlie bipolar disorder (BP). There were several neurobiological similarities between neuro-progression in BP and aging. Patients of BP also had many changes that were associated with early senescence. Meta-analysis showed that the association between dementia and BP were stronger than those with major depressive disorder, too. Therefore, some researchers proposed the theory of bipolar disorder as an illness of accelerated aging. However, BP is frequently under-recognized and misdiagnosed, especially bipolar II disorder (BP-II). Although the lifetime prevalence rate of BP-II ranges around 3-11%, many with BP-II were misdiagnosed as major depressive disorder and did not receive appropriate treatment. Therefore, neuro-progression may be found after decades of disease onset. The neuro-progression process, as accelerated aging process, may occur in the middle age period in BP-II patients, and contribute to the cognitive deficits, which were typically shown in old aged subjects with neurocognitive disorder. However, most of the past studies focused on bipolar I disorder (BP-I), there were few studies to investigate the early neuro-progression process in BP-II. Treatments for the cognitive deficits in middle-to-old aged BP-II patients were also lacked in literature.

Memantine (MM) has neuroprotective effects through the mechanisms of reducing neuroinflammation and increasing neurotrophic factors. The previous study showed that add-on low dose MM with mood stabilizers may attenuate inflammatory status and improve metabolic dysregulation in BP patients. Therefore, the investigators hypothesized that add-on MM 5 mg/day may reduce chronic inflammation, and subsequently improve neuro-progression process and cognitive function in middle-to-old aged BP-II patients. In current proposal, the investigators will conduct a randomized double-blind placebo-controlled study. The investigators will recruit 100-120 patients with BP-II who are older than 40 years old in three years, and allocate them to add-on MM or placebo plus standard valproic acid treatment in a 1: 1 ratio. The investigators will follow up the participants for 12 weeks and measure the severity of mood symptoms, neuropsychological tests and inflammatory markers to evaluate the therapeutic effects of add-on MM. The current proposal will provide the important data in whether add-on MM is able to improve the cognitive deficits due to neuro-progression in BP-II, and to prevent disease progression to a more severe form of neurocognitive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient or legal representative.
2. Male or female patient aged ≧40 years.
3. A diagnosis of bipolar II disorder according to Diagnostic and Statistical Manual of Mental Disorders criteria made by a specialist in psychiatry.
4. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

1. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study.
2. Females who are pregnant or lactation.
3. Comorbid with substance-related disorders, borderline personality disorder, schizophrenia, mental retardation, dementia or other major psychiatric disorders. But comorbid with anxiety disorder or tobacco use disorder is not an exclusion criteria.
4. Current evidence of an uncontrolled and/or clinically significant medical condition, e.g., cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation.
5. History of allergy or intolerable side effects of valproic acid, memantine, risperidone, fluoxetine, lorazepam.
6. History of receiving electroconvulsive therapy.
7. Levels of total bilirubin, aspartate aminotransferase(AST)、alanine transaminase(ALT) were elevated more than twice of normal range. Levels of Blood urea nitrogen(BUN) and creatinine were elevated more than three times of normal range.
8. Presence of alcohol abuse/dependence or illicit drug abuse/dependence in previous 6 months before beginning of study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Memory function | 12 weeks
  The participants will receive the exam of Wechsler Memory Scale-III (WMS-III) at baseline and at the endpoint (after receiving memantine or placebo treatment for 12 weeks). WMS-III composite scores were calculated for the eight standardized primary indices: Auditory Immediate (AIM, range from 50-156), Visual Immediate (VIM, range from 47-162 ), Immediate Memory (IM, range from 40-164 ), Auditory Delayed (ADM, range from 46-162), Visual Delayed (VDM, range from 43-156), Auditory Recognition Delayed (ARDM, range from 55-145), General Memory (GM, range from 40-168), and Working Memory (WM, range from 45-156 ). Higher scores indicate better performance.

SECONDARY OUTCOMES:
executive function | 12 weeks
  The participants will receive the exam of Wisconsin Card Sorting Test (WCST)at baseline and at the endpoint (after receiving memantine or placebo treatment for 12 weeks). Performance on the WCST was scored in terms of the total number of errors (TNE, range form 0-128), perseverative errors (PE, range from 0-118), conceptual level responses (CLRs, range from 0-100%), number of categories completed (NCC, range form 0-12), and trials to complete the first category (TCC, range from 0-128). Higher scores indicate worse performance in TNE, PE, and TCC. Higher scores indicate better performance in CLRs and NCC.
Attention | 12 weeks
  The participants will receive the exam of Continuous performance tests at baseline and at the endpoint (after receiving memantine or placebo treatment for 12 weeks). The CPT produces a standard set of performance measures that include the number of errors of omission and errors of commission. (1) Errors of omission occur when the participant fails to respond to the target stimulus. The omission errors t-scores are ranged from 20-80 (0-100%). Higher scores indicated worse performance. (2) Errors of commission occur when the participant responds to a non-target (X) stimulus. The commission errors t-scores are ranged from 20-80 (0-100%). Higher scores indicated worse performance.
Processing speed | 12 weeks
  The participants will receive the exam of Trial-Making Test at baseline and at the endpoint (after receiving memantine or placebo treatment for 12 weeks). Higher score indicate worse performance.
Inflammatory status | 12 weeks
  The plasma levels of cytokines and neurotrophic factors, tumor necrosis factor α (TNF-α[pg/mL]), C-reactive protein (CRP[pg/mL]), transforming growth factor β1 (TGF-β1 [pg/mL]), interleukin 6( IL-6[pg/mL]), interleukin 8(IL-8[pg/mL]), interleukin 1β (IL-1β[pg/mL]), and brain-derived neurotrophic factor(BDNF[pg/mL]), will be measured in participants at baseline and at the endpoint (after receiving memantine or placebo treatment for 12 weeks).

OTHER OUTCOMES:
Mood symptoms severity | 12 weeks
  The participants will receive the evaluation of Hamilton Depression Rating Scale (HDRS) and Young Mania Rating Scale at baseline and at the endpoint (after receiving memantine or placebo treatment for 12 weeks). The total scores of HDRS range from 0-52. The total scores of YMRS range from 0-60. Higher scores indicate more severe mood symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yun Wang, Principal Investigator — College of Medicine, National Cheng Kung University
Locations (1):
- Department of Psychiatry, National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No